CLINICAL TRIAL: NCT07268313
Title: English Title: Complete Remission Study Subtitle: Discontinuation of Mepolizumab or Dupilumab After at Least 12 Months Without Symptoms in Patients With Severe Chronic Rhinosinusitis With Polyps - a National Danish RCT Study
Brief Title: Complete Remission After Treatment With Biologics for Nasal Polyps
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kasper Aanaes, Medical doctor, phd., Principal investigator, associated professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rigshospitalet-ENT-1
Record Dates: First submitted 2025-09-02; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — dupilumab; mepolizumab

STUDY DESIGN:
Intervention Model Description: One intervention group stops treatment (but starts again if any symptom returns), one control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Continue Drug D (Active Comparator): Participants continue their usual treatment with Drug Dupi throughout the study.
  Interventions: Drug: DUPIXENT®
- Arm 2: Stop Drug D (Experimental): Participants discontinue Drug Dupi at baseline and receive no active treatment during the study.
  Interventions: Other: Dupi discontinuation
- Arm 3: Continue Drug M (Active Comparator): Participants continue their usual treatment with Drug Mepo throughout the study.
  Interventions: Drug: NUCALA®
- Arm 4: Stop Drug M (Experimental): Participants discontinue Drug Mepo at baseline and receive no active treatment during the study.
  Interventions: Other: Mepo discontinuation

INTERVENTIONS:
Drug: DUPIXENT® — Continue Dupixent
  Arms: Arm 1: Continue Drug D
Drug: NUCALA® — "Continue Nucala
  Arms: Arm 3: Continue Drug M
Other: Dupi discontinuation — Stop taking Dupixent at baseline; no substitute is given
  Arms: Arm 2: Stop Drug D
Other: Mepo discontinuation — Stop taking Nucala at baseline; no substitute is given
  Arms: Arm 4: Stop Drug M

SUMMARY:
In this RCT the investigators randomize patients who are treated with biologic treatment (Nucala or Dupixent) due to nasal polyps and have controlled disease within the last year to either stop treatment og continue as a control group.

DETAILED DESCRIPTION:
11 Protocol Synopsis 11.1. EU trial number and full trial title: 2024- 5196285-25-00 English title: Complete remission study Subtitle: Discontinuation of Mepolizumab or Dupilumab after at least 12 months without symptoms in patients with severe Chronic rhinosinusitis with polyps - a National Danish RCT study.

11.2. Rationale Specify background and hypothesis of the trial. The Danish Medicines Council has decided that well-controlled patients with nasal polyps should try to cease the medication after two years of treatment with biologics (Mepolizumab or Dupilumab). The investigators find this better to do in a RCT. Based on the experience from asthma patients this could be done in some patients without the symptoms reoccur.

11.3. Objective Specify the main and secondary objectives of the trial. The main objective is to find the percentage of patients in complete remission (no or few symptoms) who can cease the biologic treatment and keep being in remission. The secondary objective is to observe if one or the other drug is more likely to give this result.

11.4. & 11.5 Main and secondary trial endpoints: The main endpoint is to monitor the percentage of patients who do not have recurrence of their sino-nasal symptoms when they cease medicine. This is evaluated at baseline and after 12,26,38,52 weeks, however, the patients can contact the investigators at any time if symptoms reoccur. A control group is included and it is assumed that patients kept on treatment will keep being in complete remission. No adverse effects are expected, thus no new medication is started.

11.6. Trial design: Non-blinded, prospective RCT. Half the included patients will keep their treatment unchanged (control-group) the other half will stop the biological treatment (everything else unchanged). Every individual participant will have a 52-week follow-up period. If a participant in the trial group gets symptoms and feel partly uncontrolled they will start treatment again with same drug, dose and interval as before the cease.

11.7. Trial population: Patients over 18 years of age, who have been on hospital administrated biologic treatment for at least 1½ year and have been in remission for at least a year.

11.8. Interventions: The participants are randomized into two groups: one group (33 patients) will be the control group with no change in their treatment, the other group (33 patients) will cease treatment.

11.9. Ethical considerations. The investigators have very few ethical concerns by conducting this study. It is highly unlikely that any side effects will occur, thus there is no suspicion that reducing dose of biologics gives risks of side effects.

Further, none of the examinations or questionnaires are add-on to the examinations that the patients must go through when being in biologic treatment.

The investigators only concern is that some patients will experience recurrence of sino-nasal and/or asthma symptoms when stopping the biologic medicine. However, there is a plan for handling this safely. Lastly, it should also be kept in mind that the Danish medicines council recommends trying to stop the treatment, thus the investigators find it better to do this under RCT conditions.

ELIGIBILITY:
Inclusion Criteria:

5.1 Inclusion criteria (all must be fulfilled)

Inclusion criteria:

At the time when the patient started biological treatment, they must have fulfilled the EPOS criteria for initiation of biologic treatment (REF EPOS):

* Fulfil the criteria for CRSwNP
* Presence of bilateral polyps in a patient
* Had ESS (sinus surgery) (exceptional circumstances excluded)
* Fulfil at least three of the following five criteria Evidence of type 2 inflammation Need for (and treated with) systemic corticosteroids or contraindication to these SNOT-22 score of 40 or above Significant loss of smell Asthma needing regular inhaled corticosteroids

To enter this study, the patient must be:

* Above 18 years of age
* Currently be in treatment with either Dupilumab (300 mg) or Mepolizumab (100 mg) with treatment every fourth week. This treatment should have been stable/unchanged for at least three months.
* Within the latest year, the patient must at all times have scored all the below symptoms of CRS five or below on a VAS scale from 0 - 10 - Doing this, it is according to the EPOS defined as controlled disease. The items are: nasal blockage, rhinorrhea/postnasal drip, facial pain/pressure, smell, sleep disturbance or fatigue) Please view appendix 2.
* Within the latest year the nasal endoscopy cannot have showed polyp score of more than 1+1 out of 4+4, further, no thick secretions or general oedema must have been present.
* Within the latest year the patient is not allowed to have had ESS or rescue treatment for their CRSwNP (antibiotics or systemic steroids)
* The patient must be able to understand Danish and able to sign an informed content.

Exclusion Criteria:

* In the twelve months of remission the patient is not allowed to have had AECRS (acute exacerbation of chronic rhinosinusitis). A common cold is allowed.
* Polyp removal in the out-patient clinic may not have been performed within the last 3 months.
* In the twelve months of remission the patient cannot at any time have scored higher than 1.2 on the ACQ questionnaire, meaning that the patient does not have uncontrolled asthma (Appendix 3).
* Patients who, because of language barriers, are not able to understand written information and, thus, are not able to answer questionnaires.
* Patients who currently receive biologics for any other disease (asthma not included)
* Patients who are not able to give informed consent (i.e., patients who are permanently incapable)
* Patients who are not eligible because of the investigator's judgement
* Patients who experience pregnancy during the study will be excluded after an unscheduled visit (LOCF) - active IVF treatment. (Please look belove)
* Patients who have or recently have had illness, such as cancer that or its treatment is expected to significantly affect morbidity and/or quality of life in the next two years
* Unwillingness to follow the study procedure
* Hypersensitivity to any of either Dupilumab or Mepolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Enrollment: 66 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who can continue being in complete remission being out of biologic treatment. | One year observaton
  It is known that some asthma patients after years of treatment can stop taking biologics without regaining symptoms. Further, studies have shown that a lot of patients can be without symptoms taking biologics every 12th week.
  The definition of being in control, also called complete remission, is: not scoring higher than 5 (range 0 -10) on a Visual Analogue Scale (VAS) on nasal blockage, rhinorrhea, facial pressure, decreased smell or sleep; 0 being no symptoms and 10 being worst imaginable further no antibiotics, systemic steroids or surgery should be needed and the nasal examination must also be unchanged.
  The primary outcome is to observe how many, if any, patients can stop their biologic treatment still being in complete remission. This is evaluated by VAS questionnaires and nasal endoscopy every third month or even more frequent if the patient has symptoms.
  This is compared with the control group that has the same follow-up regime.

SECONDARY OUTCOMES:
Is there any difference in what drug (Dupixent or Nucala) the patient was treated with before they stopped in the ability to obtain complete remission | One year observation
  When randomizing the patients they are stratified for what drug, they are treated with - Dupixent or Nucala. If some of the patients can be out of treatment for a year, thereby obtain-ing complete remission. Thus, the secondary outcome is to describe the percentage of pa-tients with complete remission who started on Dupixent and Nucala, respectively.

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Rigshospitalet, Copenhagen, Region H
  - Nordsjællands hospital, Hillerød, Region H
  - Køge øre næse hals afd, Køge, Region Sj
  - Dept. of otorhinolaryngology, Odense, Odense, Region Syd
  - Vejle sygehus, Vejle, Region S
  - Gødstrup Hospital, Gødstrup

IPD SHARING:
Plan to Share IPD: No